CLINICAL TRIAL: NCT00258531
Title: Evaluation of 3-Dimensional Magnetic Imaging During Colonoscopy for Visualisation of Endoscope Localisation
Brief Title: Evaluation of 3-Dimensional Magnetic Imaging During Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sykehuset Telemark (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STHF Gastro 01
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2006-07-28 (Estimated); Status verified 2005-06

CONDITIONS: Any Symptom Requiring Colonoscopy

INTERVENTIONS:
Device: Olympus ScopeGuide®, 3-dimentional magnetic imager

SUMMARY:
* A commercial 3-dimentional magnetic imaging system (Olympus ScopeGuide) is available for routine use during colonoscopy.
* No randomised trials have been performed to evaluate if, and to what extent, the use of this technology may improve the coecal intubation rate and reduce the patient's experience of discomfort and pain by making the insertion of the endoscope easier

DETAILED DESCRIPTION:
Endoscopist at different level of experience are to participate. Patients routinely referred to the outpatients department for colonoscopy are asked to participate in a randomised trial where coecal intubation rate and pain experienced by the patient are end-point. Written informed consent is obtained. For each endoscopist, allocated patients are randomised to colonoscopy with no imaging technique (usual care) or using the 3-dimentional imager.

ELIGIBILITY:
Inclusion Criteria:

* A successive series of patients referred for routine colonoscopy

Exclusion Criteria:

* Age under 18 years
* Pregnant women
* Persons with pacemaker
* Unwillingness to restrict sedation to "on demand"
* Inability to understand the information given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2003-06; Study Completion 2005-06

PRIMARY OUTCOMES:
Pain experienced during colonoscopy

SECONDARY OUTCOMES:
Coecal intubation rate

CONTACTS AND LOCATIONS:
Overall Officials: Geir Hoff, MBChB PhD, Principal Investigator — Sykehuset Telemark
Locations (1):
- Medical Outpatients dept, Sykehuset Telemark, Skien, Norway